CLINICAL TRIAL: NCT07269002
Title: "Role of Clinical Pharmacy and Mobile Medical Applications in Detection and Minimization of Different Medication Errors in Hospitalized Patients From Adults and Children".
Brief Title: Clinical Pharmacist Impact Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Abd Elhamid Mohammed Tony, Clinical Pharmacist and Principal Investigator, Beni-Suef University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: F PH-BSU-HREC-0001025
Record Dates: First submitted 2025-11-21; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Medication Safety; Preventable Medication Harm; Pharmacotherapy Optimization
Keywords: Clinical pharmacist; Medication review; Smartphone clinical apps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual inpatient medication practices before implementation of the pharmacist-led safety program.
- Intervention (Other): Structured pharmacist-led medication review and safety support using smartphone clinical decision-support applications.
  Interventions: Other: Pharmacist-Led Medication Safety Program

INTERVENTIONS:
Other: Pharmacist-Led Medication Safety Program — A structured clinical pharmacist program that includes inpatient medication review, identification of potential medication-related problems, and use of smartphone-based clinical decision-support applications to support therapeutic decision-making and enhance medication safety practices.
  Arms: Intervention

SUMMARY:
This study evaluated a pharmacist-led medication-safety program in hospitalized patients. The program included routine inpatient medication review and the use of smartphone-based clinical decision-support applications to identify potential medication issues and support therapeutic decision-making. The study was conducted in both adult and pediatric inpatients as part of routine clinical care. No investigational drugs or devices were used.

DETAILED DESCRIPTION:
This study was conducted to assess the impact of a structured pharmacist-led medication-safety program implemented across inpatient units in a multispecialty hospital. The program incorporated routine clinical pharmacist review of inpatient medication therapy and the use of smartphone-based clinical decision-support applications to assist with identifying potential medication issues and supporting therapeutic optimization.

The intervention was applied prospectively in both adult and pediatric inpatients receiving pharmacologic treatment. All activities were performed as part of routine clinical service enhancement, without the use of investigational drugs or devices. The study focused on evaluating medication-safety indicators, clinical process measures, and patient-related outcomes before and after implementation of the pharmacist-led program.

The aim of the project was to enhance medication accuracy, reduce preventable medication-related problems, and support evidence-based decision-making in a real-world hospital environment. This description summarizes the overall service-improvement approach without disclosing study-specific operational details.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients receiving medication therapy

Adult and pediatric inpatients

Patients receiving at least one scheduled medication dose during admission

Exclusion Criteria:

* Patients not receiving any pharmacologic treatment

Patients admitted for procedures with no medication administration

Patients discharged before assessment could be performed

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3600 (Actual)
Dates: Start 2025-03-15 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Medication-Safety Composite Indicator | From hospital admission through study completion (an average of 5 days)
Medication-Safety Composite Indicator | From hospital admission through study completion (an average of 5 days)
  A composite measure assessing medication-safety performance in inpatient settings, including identification of medication discrepancies, potential medication risks, and pharmacist-detected issues during routine clinical care. The measure reflects overall improvement in medication-safety processes following the implementation of the pharmacist-led program.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Coordination Unit, Banī Suwayf, Egypt